CLINICAL TRIAL: NCT06249113
Title: Effectiveness of Adjuvant Continuous Lidocaine in General Anesthesia on Depth of Anesthesia (qCON), Pain Response (qNOX), and Blood Sugar Levels in Elective Primary Tumor Craniotomy Surgery
Brief Title: Effectiveness of Continous Adjuvant Lidocaine on General Anaesthesia on Tumor Craniotomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Arief Cahyadi, Anestesiologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUAnes1001
Record Dates: First submitted 2024-01-16; First posted 2024-02-08 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Surgery; Anesthesia; Functional; Haemodynamic Instability
Keywords: Adjuvant Continuous Lidocaine; General Anesthesia; Depth of Anesthesia; Pain Response; Blood Sugar Levels; Elective Primary Tumor Craniotomy Surgery
MeSH Terms: interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NaCl 0.9% continous intravenous on tumor craniotomy surgery (Placebo Comparator): NaCl 0.9% continous intravenous on general anesthesia during tumor craniotomy surgery
  Interventions: Drug: NaCl 0.9%
- Adjuvant lidocaine continous intravenous on tumor craniotomy surgery (Active Comparator): Adjuvant lidocaine continous intravenous on general anesthesia during tumor craniotomy surgery
  Interventions: Drug: Adjuvant lidocaine continous

INTERVENTIONS:
Drug: NaCl 0.9% — NaCl 0.9% continous intravenous on tumor craniotomy surgery
  Other Names: Normal Saline
  Arms: NaCl 0.9% continous intravenous on tumor craniotomy surgery
Drug: Adjuvant lidocaine continous — Adjuvant lidocaine continous intravenous on tumor craniotomy surgery
  Other Names: Lidocaine Intravenous
  Arms: Adjuvant lidocaine continous intravenous on tumor craniotomy surgery

SUMMARY:
This study aims to investigate the effect of adjuvant continuous lidocaine in General Anesthesia on Depth of Anesthesia (qCON), Pain Response (qNOX), and Blood Sugar Levels in Elective Primary Tumor Craniotomy Surgery

DETAILED DESCRIPTION:
Craniotomy for resection of brain tumors is frequently performed in neurosurgical practice. Craniotomy surgery is currently starting to use the Enhanced Recovery After Surgery (ERAS) protocol, namely for intraoperative pain management. Intraoperative pain can be evaluated through intraoperative hemodynamic conditions or can also use qCON and qNOX parameters and blood sugar levels. Perioperative pain management in the form of continuous intravenous lidocaine shows a role in reducing intraoperative pain. However, the use of intravenous lidocaine in ERAS protocols is still debated. So this study aims to use general anesthesia with continuous IV lidocaine adjuvant general anesthesia to affect depth of anesthesia (qCONtm) and intraoperative pain response in the form of values (qNOXtm), and blood sugar levels during elective primary tumor craniotomy.

The method is a Double-Blinded Randomized Control Trial. 60 patients aged 18-65 years who were diagnosed with craniotomy supratentorial tumor were randomly allocated to either Adjuvant Continuous Lidocaine (intervention group) or Normal Saline 0.9% (control group). Both drugs are given in a 20 ml syringe. The primary outcome measure of the study was the intraoperative of qCON, qNOX, and Blood Sugar. While the secondary outcome was the intraoperative hemodynamic.

All patients will be induced by general anesthesia using fentanyl 3 μg/kg IV as coinduction and propofol 1 mg/kg until the patient falls asleep. After induction, patients who receive lidocaine will receive a continuous intravenous infusion of 2 mg/kg/hour of lidocaine while other patients are given 0.9% NaCl as control. All patients data of hemodynamics, qCon, QNox, and blood glucose recorded and will be analyze.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 - 65 years with a diagnosis of brain tumor supratentorial who will undergo craniotomy by opening the dura
* ASA physical status 1-3
* Surgery using a head pin
* The level of consciousness was assessed with the Glasgow Coma Scale 15

Exclusion Criteria:

1. The patient's family or guardian refuses informed consent included in the research
2. The patient has atrioventricular block
3. There is a midline shift > 5.4 mm
4. Diagnosis of glioblastoma multiforme or metastases
5. History of allergies to drugs used in the study
6. The patient routinely consumes or is administered class of drugs adrenergic agonists or antagonists (e.g., beta blockers, α-2 agonists, vasodilator, vasoconstrictor or inotropic).
7. The patient has been regularly consuming analgesic agents for the past 2 weeks.
8. The patient has a history of cardiac arrhythmia, kidney or liver disease based on the results of the history and confirmed by further examination.
9. Suffering from diabetes mellitus or taking anti-drugs hyperglycemia based on preoperative assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Depth of Anaesthesia | Intraoperation
  Depth of Anaesthesia measured by qCON index on CONOX monitor. qCON ranges from 0 to 99. A qCON index of more than 60 indicates inadequate use of sedative agents, whereas a qCON of less than 40 indicates excessive sedation
Pain Response | Intraoperation
  Pain Response measured by qNOX index on CONOX monitor. The qNOX index uses a scale from 0 to 99 where 99 indicates a high probability of response to noxious stimulation. A decreasing index value means a smaller probability of response to the stimulus
Blood Sugar Levels | Intraoperation
  Blood Sugar Levels measured by blood test during surgery

SECONDARY OUTCOMES:
Blood Pressure | Intraoperation
  blood pressure (mm/Hg) shown on the monitor during surgery, induction, intubation, head pin installation, and skin incision, bone opening, dura mater opening, skin suturing. Blood Preasure includes systolic (mmHg), Diastolic (mmHg), and Mean Arterial Pressure (mmHg)
Heart Rate | Intraoperation
  Heart Rate (times/minutes) shown on the monitor during surgery, induction, intubation, head pin installation, and skin incision, bone opening, dura mater opening, skin suturing
Body Temperature | Intraoperation
  Body Temperature (celsius) shown on the monitor during surgery, induction, intubation, head pin installation, and skin incision, bone opening, dura mater opening, skin suturing

CONTACTS AND LOCATIONS:
Overall Officials: Arief Cahyadi, Specialist, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Robles P, Fiest KM, Frolkis AD, Pringsheim T, Atta C, St Germaine-Smith C, Day L, Lam D, Jette N. The worldwide incidence and prevalence of primary brain tumors: a systematic review and meta-analysis. Neuro Oncol. 2015 Jun;17(6):776-83. doi: 10.1093/neuonc/nou283. Epub 2014 Oct 13. PMID 25313193
- [Background] Dashti M, Amini S, Azarfarin R, Totonchi Z, Hatami M. Hemodynamic changes following endotracheal intubation with glidescope((R)) video-laryngoscope in patients with untreated hypertension. Res Cardiovasc Med. 2014 May;3(2):e17598. doi: 10.5812/cardiovascmed.17598. Epub 2014 Apr 1. PMID 25478537
- [Background] Can BO, Bilgin H. Effects of scalp block with bupivacaine versus levobupivacaine on haemodynamic response to head pinning and comparative efficacies in postoperative analgesia: A randomized controlled trial. J Int Med Res. 2017 Apr;45(2):439-450. doi: 10.1177/0300060516665752. Epub 2017 Mar 7. PMID 28415943
- [Background] Greisen J, Juhl CB, Grofte T, Vilstrup H, Jensen TS, Schmitz O. Acute pain induces insulin resistance in humans. Anesthesiology. 2001 Sep;95(3):578-84. doi: 10.1097/00000542-200109000-00007. PMID 11575527
- [Background] Marik PE, Bellomo R. Stress hyperglycemia: an essential survival response! Crit Care. 2013 Mar 6;17(2):305. doi: 10.1186/cc12514. PMID 23470218
- [Background] Gruenbaum SE, Meng L, Bilotta F. Recent trends in the anesthetic management of craniotomy for supratentorial tumor resection. Curr Opin Anaesthesiol. 2016 Oct;29(5):552-7. doi: 10.1097/ACO.0000000000000365. PMID 27285727
- [Background] Beaussier M, Delbos A, Maurice-Szamburski A, Ecoffey C, Mercadal L. Perioperative Use of Intravenous Lidocaine. Drugs. 2018 Aug;78(12):1229-1246. doi: 10.1007/s40265-018-0955-x. PMID 30117019
- [Background] McKay A, Gottschalk A, Ploppa A, Durieux ME, Groves DS. Systemic lidocaine decreased the perioperative opioid analgesic requirements but failed to reduce discharge time after ambulatory surgery. Anesth Analg. 2009 Dec;109(6):1805-8. doi: 10.1213/ANE.0b013e3181be371b. PMID 19923506
- [Background] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Background] Peng Y, Zhang W, Kass IS, Han R. Lidocaine Reduces Acute Postoperative Pain After Supratentorial Tumor Surgery in the PACU: A Secondary Finding From a Randomized, Controlled Trial. J Neurosurg Anesthesiol. 2016 Oct;28(4):309-15. doi: 10.1097/ANA.0000000000000230. PMID 26397235
- [Background] Hani U, Bakhshi SK, Shamim MS. Enhanced Recovery after Elective Craniotomy for Brain Tumours. J Pak Med Assoc. 2019 May;69(5):749-751. PMID 31105305
- [Background] Lapointe S, Perry A, Butowski NA. Primary brain tumours in adults. Lancet. 2018 Aug 4;392(10145):432-446. doi: 10.1016/S0140-6736(18)30990-5. Epub 2018 Jul 27. PMID 30060998
- [Background] Kirby S, Purdy RA. Headaches and brain tumors. Neurol Clin. 2014 May;32(2):423-32. doi: 10.1016/j.ncl.2013.11.006. Epub 2013 Dec 27. PMID 24703537
- [Background] Vacas S, Van de Wiele B. Designing a pain management protocol for craniotomy: A narrative review and consideration of promising practices. Surg Neurol Int. 2017 Dec 6;8:291. doi: 10.4103/sni.sni_301_17. eCollection 2017. PMID 29285407
- [Background] Chowdhury T, Garg R, Sheshadri V, Venkatraghavan L, Bergese SD, Cappellani RB, Schaller B. Perioperative Factors Contributing the Post-Craniotomy Pain: A Synthesis of Concepts. Front Med (Lausanne). 2017 Mar 1;4:23. doi: 10.3389/fmed.2017.00023. eCollection 2017. PMID 28299313
- [Background] Yam MF, Loh YC, Tan CS, Khadijah Adam S, Abdul Manan N, Basir R. General Pathways of Pain Sensation and the Major Neurotransmitters Involved in Pain Regulation. Int J Mol Sci. 2018 Jul 24;19(8):2164. doi: 10.3390/ijms19082164. PMID 30042373
- [Background] Melia U, Gabarron E, Agusti M, Souto N, Pineda P, Fontanet J, Vallverdu M, Jensen EW, Gambus P. Comparison of the qCON and qNOX indices for the assessment of unconsciousness level and noxious stimulation response during surgery. J Clin Monit Comput. 2017 Dec;31(6):1273-1281. doi: 10.1007/s10877-016-9948-z. Epub 2016 Oct 20. PMID 27766525
- [Background] Jensen EW, Valencia JF, Lopez A, Anglada T, Agusti M, Ramos Y, Serra R, Jospin M, Pineda P, Gambus P. Monitoring hypnotic effect and nociception with two EEG-derived indices, qCON and qNOX, during general anaesthesia. Acta Anaesthesiol Scand. 2014 Sep;58(8):933-41. doi: 10.1111/aas.12359. Epub 2014 Jul 4. PMID 24995461
- [Background] Muller JN, Kreuzer M, Garcia PS, Schneider G, Hautmann H. Monitoring depth of sedation: evaluating the agreement between the Bispectral Index, qCON and the Entropy Module's State Entropy during flexible bronchoscopy. Minerva Anestesiol. 2017 Jun;83(6):563-573. doi: 10.23736/S0375-9393.17.11262-9. Epub 2017 Feb 8. PMID 28177205
- [Background] Jensen EW. New findings and trends for depth of anesthesia monitoring. Korean J Anesthesiol. 2018 Oct;71(5):343-344. doi: 10.4097/kja.d.18.00277. Epub 2018 Oct 1. No abstract available. PMID 30301320
- [Background] Christenson C, Martinez-Vazquez P, Breidenstein M, Farhang B, Mathews J, Melia U, Jensen EW, Mathews D. Comparison of the Conox (qCON) and Sedline (PSI) depth of anaesthesia indices to predict the hypnotic effect during desflurane general anaesthesia with ketamine. J Clin Monit Comput. 2021 Dec;35(6):1421-1428. doi: 10.1007/s10877-020-00619-3. Epub 2020 Nov 19. PMID 33211251
- [Background] Hermanns H, Hollmann MW, Stevens MF, Lirk P, Brandenburger T, Piegeler T, Werdehausen R. Molecular mechanisms of action of systemic lidocaine in acute and chronic pain: a narrative review. Br J Anaesth. 2019 Sep;123(3):335-349. doi: 10.1016/j.bja.2019.06.014. Epub 2019 Jul 11. PMID 31303268
- [Background] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177
- [Background] Nakhli MS, Kahloul M, Guizani T, Zedini C, Chaouch A, Naija W. Intravenous lidocaine as adjuvant to general anesthesia in renal surgery. Libyan J Med. 2018 Dec;13(1):1433418. doi: 10.1080/19932820.2018.1433418. PMID 29433385
- [Background] Gaughen CM, Durieux M. The effect of too much intravenous lidocaine on bispectral index. Anesth Analg. 2006 Dec;103(6):1464-5. doi: 10.1213/01.ane.0000247700.71278.70. PMID 17122224
- [Background] Soleimanpour H, Hassanzadeh K, Vaezi H, Golzari SE, Esfanjani RM, Soleimanpour M. Effectiveness of intravenous lidocaine versus intravenous morphine for patients with renal colic in the emergency department. BMC Urol. 2012 May 4;12:13. doi: 10.1186/1471-2490-12-13. PMID 22559856
- [Background] Kandil E, Melikman E, Adinoff B. Lidocaine Infusion: A Promising Therapeutic Approach for Chronic Pain. J Anesth Clin Res. 2017 Jan;8(1):697. doi: 10.4172/2155-6148.1000697. Epub 2017 Jan 11. PMID 28239510
- [Background] DeVon HA, Piano MR, Rosenfeld AG, Hoppensteadt DA. The association of pain with protein inflammatory biomarkers: a review of the literature. Nurs Res. 2014 Jan-Feb;63(1):51-62. doi: 10.1097/NNR.0000000000000013. PMID 24335913
- [Result] Saito J, Masters J, Hirota K, Ma D. Anesthesia and brain tumor surgery: technical considerations based on current research evidence. Curr Opin Anaesthesiol. 2019 Oct;32(5):553-562. doi: 10.1097/ACO.0000000000000749. PMID 31145197
- See also: Neuro-anesthetic Management of Craniotomy-surgery in Removal Tumor Multiple Meningioma Patients: A Case Report — http://oamjms.eu/index.php/mjms/article/view/6371
- See also: Effects of indexes of consciousness (IoC1 and IoC2) monitoring on remifentanil dosage in modified radical mastectomy: a randomized trial — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4810508/
- See also: Acute stress-induced changes in hormone and lipid levels in mouse plasma — http://www.agriculturejournals.cz/pdfs/vet/2016/02/01.pdf
- See also: Efek Pemberian Lidokain Intravena Kontinu Intraoperasi terhadap Kebutuhan Isofluran dan Pemakaian Fentanil pada Operasi Dekompresi dan Stabilisasi Posterior Vertebra — http://macc.perdatin.org/index.php/my-journal/article/view/208